CLINICAL TRIAL: NCT02235103
Title: The Predictive Value of the Sperm Chromatin Dispersion Test, Halosperm®, Before and After Sperm Preparation for Clinical Pregnancy in Cases of Unexplained Infertility Treated With Intra-uterine Insemination (First Cycle) and Ovulation Induction With Clomiphene Citrate.
Acronym: DNAFRAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201316616
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Unexplained Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sperm samples

GROUPS / COHORTS (2):
- Clinical Pregnancy: Patients who are clinically pregnant after first treatment cycle with intra-uterine insemination.
  Interventions: Other: Sperm Chromatin Dispersion Test
- No Clinical Pregnancy: Patients who are not clinically pregnant after first treatment cycle with intra-uterine insemination.
  Interventions: Other: Sperm Chromatin Dispersion Test

INTERVENTIONS:
Other: Sperm Chromatin Dispersion Test
  Other Names: Halosperm®

SUMMARY:
Recent research has revealed that subtle abnormalities can be found in sperm samples that seem to be normal with conventional analysis techniques. The DNA in the sperm heads is sometimes fragmented and this may be the reason why couples with a diagnosis of unexplained infertility do not achieve pregnancy.

We are planning a study to examine the incidence of DNA fragmentation in the sperm of couples with previously unexplained infertility. In a first treatment cycle with intra-uterine insemination the percentage of DNA fragmentation in sperm will be measured. Afterwards the results of the patients who are pregnant will be compared with those of the not pregnant ones. We expect to find differences between both groups.

100 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility, i.e. female patients with ovulatory cycles and patent tubes; normal sperm analysis (WHO criteria).
* Patient agrees to have a first treatment cycle with intra-uterine insemination and ovulation-induction with clomiphene citrate.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with unexplained fertility treated with intra-uterine insemination (first cycle) and ovulation induction with clomiphene citrate.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 2 1/2 weeks after insemination
  Ultrasound to diagnose intra-uterine pregnancy

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 20 weeks after insemination
  Ultrasound to diagnose an evolutive pregnancy.
Live birth rate | 42 weeks after insemination
  Clinical report of the delivery by the obstetrician

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vandekerckhove, MD, Principal Investigator — Fertility Centre, University Hospital Ghent
Locations (1):
- Fertility Centre of the University Hospital, Ghent, East Flanders, Belgium